CLINICAL TRIAL: NCT01935947
Title: A Randomized Phase II Trial of Cytotoxic Chemotherapy With or Without Epigenetic Priming in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Azacitidine and Entinostat Before Chemotherapy in Treating Patients With Advanced Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00949; NCI-2013-00949 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NA_00081948/J1309; NA_00081948; 9253 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); 9253 (Other: CTEP); P30CA006973 (NIH); NCT01846897 (obsolete NCT alias)
Record Dates: First submitted 2013-09-03; First posted 2013-09-05 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-06

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Azacitidine; Docetaxel; entinostat; Gemcitabine; Irinotecan; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (azacitidine, entinostat, chemotherapy) (Experimental): Patients receive azacitidine SC on days 1-6 and 8-10 and entinostat PO on days 3 and 10. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or progressive disease receive chemotherapy of the treating oncologist's choice comprising irinotecan hydrochloride IV on day 1, docetaxel IV on day 1, pemetrexed disodium IV on day 1, or gemcitabine hydrochloride IV on days 1 and 8. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Docetaxel; Drug: Entinostat; Drug: Gemcitabine Hydrochloride; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Pemetrexed Disodium
- Arm II (azacitidine, entinostat, chemotherapy) (Experimental): Patients receive azacitidine PO on days 1-21 and entinostat PO on days 3 and 10. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or progressive disease receive chemotherapy of the treating oncologist's choice as in Arm A.
  Interventions: Drug: Azacitidine; Drug: Docetaxel; Drug: Entinostat; Drug: Gemcitabine Hydrochloride; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Pemetrexed Disodium
- Arm III (chemotherapy) (Active Comparator): Patients receive chemotherapy of the treating oncologist's choice as in Arm A.
  Interventions: Drug: Docetaxel; Drug: Gemcitabine Hydrochloride; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Pemetrexed Disodium

INTERVENTIONS:
Drug: Azacitidine — Given SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: Arm I (azacitidine, entinostat, chemotherapy)
Drug: Azacitidine — Given PO
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: Arm II (azacitidine, entinostat, chemotherapy)
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Drug: Entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; MS 27-275; MS-275; SNDX-275
  Arms: Arm I (azacitidine, entinostat, chemotherapy); Arm II (azacitidine, entinostat, chemotherapy)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; U-101440E
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt

SUMMARY:
This randomized phase II trial studies how well azacitidine and entinostat before chemotherapy works in treating patients with non-small cell lung cancer that has spread to other places in the body. Drugs used in chemotherapy, such as azacitidine, irinotecan hydrochloride, gemcitabine hydrochloride, docetaxel, and pemetrexed disodium, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Entinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving azacitidine and entinostat before chemotherapy may work better in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Percentage of patients progression-free at 6 months from time of randomization.

SECONDARY OBJECTIVES:

I. Progression-free survival (PFS). II. Overall survival (OS).

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM A: Patients receive azacitidine subcutaneously (SC) on days 1-6 and 8-10 and entinostat orally (PO) on days 3 and 10. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or progressive disease receive chemotherapy of the treating oncologist's choice comprising irinotecan hydrochloride intravenously (IV) on day 1, docetaxel IV on day 1, pemetrexed disodium IV on day 1, or gemcitabine hydrochloride IV on days 1 and 8. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive azacitidine PO on days 1-21 and entinostat PO on days 3 and 10. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or progressive disease receive chemotherapy of the treating oncologist's choice as in Arm A.

ARM C: Patients receive chemotherapy of the treating oncologist's choice as in Arm A.

After completion of treatment, patients are followed up every 3-6 months for 24 months and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically proven non-small cell lung cancer; tumor tissue must be available from all patients prior to initiation of protocol therapy, either from original diagnostic biopsy, or biopsy performed prior to initiation of protocol therapy
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Patients must have received 1 prior platinum containing doublet regardless of mutation status
* Patients with targetable mutation i.e. epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK), must have been treated with at least 1 prior tyrosine kinase inhibitor (TKI)
* Prior immunotherapy is allowed
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Karnofsky >= 70%)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transferase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transferase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who are receiving any other investigational agents
* Patients with uncontrolled brain metastases; patients with brain metastases must have stable neurologic status following local therapy (surgery or radiation) for at least 4 weeks, and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; patients may be treated with steroids as clinically indicated
* Patients with liver metastases that replace greater than 30% of the liver parenchyma
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to entinostat, azacitidine, mannitol, irinotecan, docetaxel, pemetrexed, or gemcitabine, or other agents used in the study
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, New York Heart Association (NYHA) class 3-4 congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated on this protocol
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-05; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Brahmer, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (5):
- United States (5):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Medical University of South Carolina, Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were seven screen failures.
Groups:
- Arm I (Azacitidine, Entinostat, Chemotherapy): Patients receive azacitidine SC on days 1-6 and 8-10 and entinostat PO on days 3 and 10. Treatment repeats every 28 days for 2 courses, then chemotherapy. Treatment repeats every 21 days.
- Arm II (Azacitidine, Entinostat, Chemotherapy): Patients receive azacitidine PO on days 1-21 and entinostat PO on days 3 and 10. Treatment repeats every 28 days for 2 courses. Patients receive chemotherapy of the treating oncologist's choice as in Arm A.
Period: Overall Study
Arm/Group | Arm I (Azacitidine, Entinostat, Chemotherapy) | Arm II (Azacitidine, Entinostat, Chemotherapy) | Arm III (Chemotherapy)
Started | 4 | 4 | 2
Epigenetic Therapy | 4 | 4 | 0
Cytotoxic Therapy | 3 | 3 | 2
Completed | 1 | 0 | 0
Not Completed | 3 | 4 | 2
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Diease Progression | 2 | 2 | 2
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Azacitidine, Entinostat, Chemotherapy): Patients receive azacitidine SC on days 1-6 and 8-10 and entinostat PO on days 3 and 10. Treatment repeats every 28 days for 2 courses then patients receive chemotherapy. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
- Arm II (Azacitidine, Entinostat, Chemotherapy): Patients receive azacitidine PO on days 1-21 and entinostat PO on days 3 and 10. Treatment repeats every 28 days for 2 courses, and then patients receive chemotherapy as in Arm A.
- Total: Total of all reporting groups
Arm/Group | Arm I (Azacitidine, Entinostat, Chemotherapy) | Arm II (Azacitidine, Entinostat, Chemotherapy) | Arm III (Chemotherapy) | Total
Number analyzed (Participants) | 4 | 4 | 2 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 2 | 5
  >=65 years | 3 | 2 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (12.6) | 62 (8.4) | 54 (2.0) | 60 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 0 | 3
  Male | 4 | 1 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 3 | 2 | 1 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Progression-free at 6 Months From the Time of Randomization
Description: The final analysis will be by Fisher's Exact test, with percentage of patients who have not progressed as the outcome variable. Using Fisher's Exact test for analysis with 55 patients per treatment group will provide 88% power to detect an increase from 40% (chemotherapy alone) to 65% (epigenetic therapy followed by chemotherapy) in the number of patients who are progression free at six months.
Time Frame: At 6 months
Population: Data was not collected to assess this outcome measure due to early study termination.
Arm/Group | Arm I (Azacitidine, Entinostat, Chemotherapy) | Arm II (Azacitidine, Entinostat, Chemotherapy) | Arm III (Chemotherapy)
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Overall Survival (OS)
Time Frame: From the time of enrollment to trial until death, assessed up to 2 years
Population: Data was not collected to assess this outcome measure due to early study termination.
Arm/Group | Arm I (Azacitidine, Entinostat, Chemotherapy) | Arm II (Azacitidine, Entinostat, Chemotherapy) | Arm III (Chemotherapy)
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Progression Free Survival
Description: From the time of randomization until radiologic or clinical progression is noted, assessed up to 2 years.
Time Frame: up to 2 years
Population: Data was not collected to assess this outcome measure due to early study termination.
Arm/Group | Arm I (Azacitidine, Entinostat, Chemotherapy) | Arm II (Azacitidine, Entinostat, Chemotherapy) | Arm III (Chemotherapy)
Number analyzed (Participants) | 0 | 0 | 0

4. Other Pre Specified Outcome: Genome-wide Techniques, Including Expression Array and Methylation Array
Description: Expression array and methylation array will be compared to response.
Time Frame: After 1 month of therapy
Population: Data was not collected to assess this outcome measure due to early study termination.
Arm/Group | Arm I (Azacitidine, Entinostat, Chemotherapy) | Arm II (Azacitidine, Entinostat, Chemotherapy) | Arm III (Chemotherapy)
Number analyzed (Participants) | 0 | 0 | 0

5. Other Pre Specified Outcome: Predictive and Prognostic Value of the Previously Defined Epigenetic Signature, Comprised of Promoter Methylation Analysis of 4 Target Genes
Time Frame: After 1 month of therapy
Population: Data was not collected to assess this outcome measure due to early study termination.
Arm/Group | Arm I (Azacitidine, Entinostat, Chemotherapy) | Arm II (Azacitidine, Entinostat, Chemotherapy) | Arm III (Chemotherapy)
Number analyzed (Participants) | 0 | 0 | 0

6. Other Pre Specified Outcome: Response to Therapy Compared to Genetic and Epigenetic Factors and Tested for Association
Time Frame: After 1 month of therapy
Population: Data was not collected to assess this outcome measure due to early study termination.
Arm/Group | Arm I (Azacitidine, Entinostat, Chemotherapy) | Arm II (Azacitidine, Entinostat, Chemotherapy) | Arm III (Chemotherapy)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 2 years
Description: Adverse events and serious adverse events will be collected for up to 30 days after the last administration of the investigational agent/intervention
Groups:
- Arm I (Azacitidine, Entinostat, Chemotherapy): Patients receive azacitidine SC on days 1-6 and 8-10 and entinostat PO on days 3 and 10. Treatment repeats every 28 days for 2 course, and then receive chemotherapy. Treatment repeats every 21 days.
- Arm II (Azacitidine, Entinostat, Chemotherapy): Patients receive azacitidine PO on days 1-21 and entinostat PO on days 3 and 10. Treatment repeats every 28 days for 2 courses, and then receive chemotherapy as in Arm A.
- Arm III (Chemotherapy): Patients receive chemotherapy as in Arm A.
Arm/Group | Arm I (Azacitidine, Entinostat, Chemotherapy) | Arm II (Azacitidine, Entinostat, Chemotherapy) | Arm III (Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/4 | 4/4 | 1/2
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Azacitidine, Entinostat, Chemotherapy) (N=4) | Arm II (Azacitidine, Entinostat, Chemotherapy) (N=4) | Arm III (Chemotherapy) (N=2)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal Cord Depression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Azacitidine, Entinostat, Chemotherapy) (N=4) | Arm II (Azacitidine, Entinostat, Chemotherapy) (N=4) | Arm III (Chemotherapy) (N=2)
anemia (Blood and lymphatic system disorders) | 2 (4) | 2 (2) | 1 (2)
AST increased (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (2) | 1 (1) | 1 (1)
Dyspnea (General disorders) | 4 (4) | 1 (1) | 1 (2)
Fatigue (General disorders) | 2 (4) | 3 (8) | 1 (11)

LIMITATIONS AND CAVEATS:
Low recruitment lead to slow accrual. Not having enough patients on the trial and high disease progression lead to closing the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT01935947/Prot_SAP_000.pdf